CLINICAL TRIAL: NCT03494075
Title: MyPaTH Story Booth
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kathleen McTigue, Professor, University of Pittsburgh
Other Study IDs: STUDY20110315
Record Dates: First submitted 2017-08-23; First posted 2018-04-11 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Narrative Medicine
Keywords: Patients; Caregivers
MeSH Terms: conditions — Narrative Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The MyPaTH Story Booth will use an (audio) "document" approach to elicit in depth experiential knowledge or perspectives from patients and caregivers by recording their personal stories.

DETAILED DESCRIPTION:
Modeled after the Storycorps project and healthtalk.org, MyPaTH Story Booth will use an (audio) "document" approach to elicit in depth experiential knowledge or perspectives from patients and caregivers by recording their personal stories. Narratives provide a powerful framework for understanding patient problems and the larger process of illness, coping, and seeking health care. Narratives can provide meaning, context, and perspective for patients' situations and insight into failures in health care delivery, particularly for marginalized patients. MyPaTH Story Booth will provide simple instructions for how participants can work with an interview partner (e.g., a family member or friend) to record their story. MyPath Story Booth may be launched sequentially at each PaTH site to establish an initial archive of patient and caregiver narratives. Individuals who record narratives will be asked to provide limited "tags" to populate a searchable database (e.g., their age, sex, interview topic). The audio booth and procedures will also be made available to PaTH affiliated researchers who wish to augment the narrative database with narratives of patient partners from specific study populations.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18

Exclusion Criteria:

* Researchers will exclude individuals who are not 18 years of age or older and/or do not provide informed consent

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anyone over the age of 18 who can provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-03; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of stories collected | September 2018
  The goal of the project is to generate a searchable archive of patient and caregiver narratives

SECONDARY OUTCOMES:
Comparison of approaches to categorize story contents | Cross-sectional analysis of the first 100 stories, September 2018
  Researchers will compare how story contents are categorized using (a) qualitative research coding with survey data collected from (b) participants and (c) study staff
Number of researchers who access the online story archive | Annually at 2 and 3 years of follow-up the number of researchers who accessed stories will be reviewed.
  To support health researchers' use of patient and caregiver narratives in formulating research questions
Number of research teams who engage stakeholders through the project | Annually at 2 and 3 years of follow-up
  The project aims to facilitate connections between individuals who have real-world insights and experience with health care or health care delivery and health researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M McTigue, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamm M, Wilson JD, Lee YJ, Norman N, Winstanley EL, McTigue KM. Substance use as subtext to health narratives: Identifying opportunities for improving care from community member perspectives. Patient Educ Couns. 2024 Nov;128:108384. doi: 10.1016/j.pec.2024.108384. Epub 2024 Aug 9. PMID 39168050
- [Background] Shah VK, Hamm M, Glynn NW, Rockette-Wagner B, McTigue K. Comparing survey data to qualitative themes in patient stories to help researchers better identify pressing community healthcare needs. J Eval Clin Pract. 2023 Aug;29(5):793-801. doi: 10.1111/jep.13837. Epub 2023 Mar 24. PMID 36961380
- [Background] McTigue KM, Fear D, Hunter K, Karanam S, Uhrig J, Alston T, Dillon S, Faust J, Kim J, LaRosa A, Postol B, Umegbolu S, Hamm M. The development of a patient and caregiver narrative archive to support patient-centered research. Eur J Pers Cent Healthc. 2018 Dec;6(4):565-570. doi: 10.5750/ejpch.v6i4.1546